

# Clinical Investigation Plan:

| Document<br>No. | Rev | Document Title (must be the same as Database/ hardcopy) | Category-<br>Folder<br>(e.g. DHF) | Folder<br>No. | Folder<br>Tab<br>section |
|---|---|---|---|---|---|
| CIA-176 | В | Clinical Investigation Plan: | CIA | 176 | 2.4 |
| Additional co | pies to: | | | | |
| Additional | Notes: | | | | |

| Ethics approval date | 21 June 2016 |
|----------------------|--------------|
| NCT number | NCT02809859 |

# **Review and Approval**

| Please tick if task complete: | Pre-release database done □, File(s) in DRAFT & Closed □ |
|---|---|
| Irene Cheung | |
| Author | |

# **Table of Contents**

| 1. | Revision | History | 4 |
|----|------------|--------------------------------------------------|----|
| 2. | List of Al | bbreviations | 4 |
| 3. | Documer | nt Information | 4 |
| | 3.1. F | Purpose and Scope | 4 |
| | | Confidentiality Statement | |
| | 3.3. F | Persons Authorized to Amend the CIP | 4 |
| | 3.4. N | Monitoring Arrangements | 4 |
| | 3.5. | Data Management | 5 |
| 4. | Investiga | tor Information | 5 |
| | 4.1. 5 | Study Principle Investigator | 5 |
| | 4.1. | 1. Co-ordinating Investigator | 5 |
| | 4.2. I | nvestigators | 5 |
| | 4.2. | 1. Co-ordinating Investigator | 5 |
| | 4.3 I | nvestigators | 5 |
| | | 1. Co-ordinating Investigator | |
| | | nvestigators | |
| | 4.4.2 | 2. Co-ordinating Investigator | 6 |
| | | Other Investigators | |
| | 4.6. I | nstitution | 6 |
| 5. | Sponsor | Information | 7 |
| | 5.1. F | Primary Sponsor Details | 7 |
| 6. | Device In | nformation | 7 |
| | 6.1. I | dentification of the Medical Device | 7 |
| | 6.2. | Device Risk Analysis and Management | 8 |
| 7. | Justificat | tion for a Clinical Trial | 8 |
| | 7.1. 5 | Synopsis | 8 |
| | 7.2. L | iterature Review | 9 |
| | 7.3. F | Preclinical Testing | 9 |
| | | Previous Clinical Experience | |
| | 7.5. J | Justification for Administration | 10 |
| 8. | Objective | es of the Clinical Investigation | 10 |
| | 8.1. H | Hypothesis | 10 |
| | | Objectives | |
| | | Population | |
| | | Risks | |
| | | Essential Requirements of the Relevant Directive | |
| 9. | | nvestigation Design | |
| | | Гуре of Investigation | |
| | | Controls | |
| | | Bias | |
| | 9.4. E | End Points | 11 |

| | 9.4.1. Primary Outcomes | 11 |
|-----|---------------------------------------------|----|
| | 9.4.2. Secondary Outcomes | 11 |
| | 9.5. Variables | 11 |
| | 9.6. Measurements | |
| | 9.7. Equipment | 12 |
| | 9.8. Inclusion / Exclusion criteria | 12 |
| | 9.9. Point of Enrolment | 13 |
| | 9.10. Patient Procedure | |
| | 9.11. Withdrawal Criteria | 14 |
| | 9.12. Number of Trial Subjects | |
| | 9.13. Follow up Plan | |
| | 9.14. Foreseeable Complications | |
| 10. | Clinical Trial Documentation | |
| | 10.1. Consent and Recruitment | |
| | 10.2. Case Report Form | |
| | 10.2.1. Case Report Form Signatories | |
| | 10.3. Insurance Statement | 15 |
| | 10.4. Record of Deviations | 16 |
| STA | TISTICAL CONSIDERATIONS | 16 |
| | 10.5. Description of the Statistical Design | 16 |
| | 10.6. Sample Size | 16 |
| | 10.7. Pass/Fail Criteria | 16 |
| | 10.8. Statistical Termination | |
| | 10.9. Statistical Procedure Deviations | |
| | 10.10. Selection Criteria | |
| | 10.11. Statistical Data Management | |
| 11. | Adverse Events and Termination | 17 |
| | 11.1. Emergency Contact Details | |
| | 11.2. Foreseeable Adverse Events | |
| | 11.3. Reporting Adverse Events | |
| | 11.4. Early Termination | |
| | 11.4.1. Investigator | 18 |
| | 11.4.2. Sponsor | 19 |
| | 11.4.3. Institutional Review Board (IRB) | 19 |
| 12. | Publication Policy | 19 |
| 13. | Approval | 19 |
| 14. | References | 19 |

| Fisher & Paykel | Clinical Investigation Plan | | |
|-----------------|-----------------------------|-----------|--------------|
| Clinical Inc | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIV | restigation Fian. | Revision: | В |

1. Revision History

| Revision | Author | Date | Description of change |
|---|---|---|---|
| Α | Irene Cheung | 12 April 2016 | First release |
| В | Irene Cheung | 21 June 2016 | Administrative changes to the questionnaire in Appendix A and B Changed sponsor contact person to Hanie Yee (Clinical Research Manager) |
| | | | Changed reporting of adverse events to Hanie Yee (Clinical Research Manager) |

### 2. List of Abbreviations

AutoCPAP Auto-adjusting Continuous Positive Airway Pressure

CIP Clinical Investigation Plan

CPAP Continuous Positive Airway Pressure

CRF Case Report Form

FPH Fisher & Paykel Healthcare

HIPPA Health Insurance Portability and Accountability Act

IB Investigator's Brochure
IRB Institutional Review Board
OSA Obstructive Sleep Apnea

### 3. Document Information

### 3.1. Purpose and Scope

This clinical investigation plan (CIP) is compiled by the investigators and sponsor (Fisher & Paykel Healthcare (FPH)). The CIP is designed to optimize the scientific validity and reproducibility of the results of this study in accordance with current clinical knowledge and practice so as to fulfil the objectives of the investigation. The investigator and the sponsor will store the current copy and all previous copies of the CIP.

The purpose of the clinical investigation, Section 8 Objectives of the Clinical Investigation.

### 3.2. Confidentiality Statement

This document contains confidential information belonging to Fisher & Paykel Healthcare and is provided for the sole purpose of enabling an evaluation of a possible collaboration with Fisher & Paykel Healthcare to undertake the proposed clinical research. This document must be maintained in a confidential manner at all times and any disclosure, distribution or reproduction of this document outside the intended purpose is prohibited.

### 3.3. Persons Authorized to Amend the CIP

### 3.4. Monitoring Arrangements

| Fisher & Paykel | Clinical Investigation Plan | | | |
|-----------------|-----------------------------|---|-----------|--------------|
| Clinical Inc | rectigation Plan: | | Doc. No: | CIA No: 176 |
| Cimicai inv | restigation Plan: | R | Revision: | В |



The details can be found in the monitoring plan.

# 3.5. Data Management

# 4. Investigator Information

# 4.1. Study Principle Investigator

Name: Matt Uhles

Address: Clayton Sleep Institute Email: uhlesm@claytonsleep.com

Phone: 314-645-6005

### 4.1.1. Co-ordinating Investigator

Name: Angela Lindsey

Address: Clayton Sleep Institute Email: LindseyA@claytonsleep.com

Phone: 314-645-6005

# 4.2. Investigators

### 4.2.1. Co-ordinating Investigator

# 4.3. Investigators

| Fishe | er&Paykel LTHCARE Clinical Investigation Plan | | |
|---|---|---|---|
| | Clinical Investigation Plan: | Doc. No: | CIA No: 176 |
| | Chinical hivestigation I fain. | Revision: | В |
| | 40.4 On andication locations | | |
| | 4.3.1. Co-ordinating Investigator | | |
| 1.4. | Investigators | | |
| | 4.4.1. Co-ordinating Investigator | | |
| | 4.4.1. 00 ordinating invostigator | | |
| | 4.4.2. Co-ordinating Investigator | | |
| <b>1.5.</b> | Other Investigators | | |
| 1.6. | Institution | | |

| Fisher | & Paykel<br>HCARE | Clinical Investigation Plan | | |
|---|---|---|---|---|
| | CI II II II | N | Doc. No: | CIA No: 176 |
| | Clinical Investigation | n Plan: | Revision: | В |
| _ | 0 | | | |
| 5. | Sponsor Info | rmation | | |
| 5.1. | <b>Primary Sponso</b> | or Details | | |
| √ame | of Business: Fisher | & Paykel Healthcare Limited | | |
| | | kel Place, East Tamaki, Auckland, New Zealand. | | |
| <b>3</b> . | <b>Device Inform</b> | nation | | |
| 5.1. | identification of | the Medical Device | | |
| Γla :.a | timational doub | | . 4. 46 | |
| | | e will provide continuous positive airway pressure | e to the pa | irticipant via a |
| reatn | ing tube and interfa | ice (mask). | | |

| Fisher & Paykel<br>HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Invo | estigation Plans | Doc. No: | CIA No: 176 |
| Clinical inve | stigation Plan: | Revision: | В |
| 6.2. Device Ris | sk Analysis and Management | | |
| | devices used in this clinical investigation will | undergo device rist | k analysis an |
| _ | o being released for clinical investigation. Eviden | _ | - |
| • | linical Investigation Folder (CIA-176). | oo or are new manag | omoni proces |
| | , | | |
| All contraindications | s, warnings, precautions and adverse effects of u | ising this device are | included in th |
| device manuals, file | ed in CIA-176, | | |
| - | se events or adverse device effects will be inc | | _ |
| -older (CIA-176), ti | ne site regulatory file and reported on the particip | pant's case report to | rm (CRF). |
| 7. Justifica | tion for a Clinical Trial | | |
| | non for a Chilical Thai | | |
| 7.1. Synopsis | CDAD upor will be recruited into this | atudy to avalue | ata tha alinia |
| erformance | e CPAP users will be recruited into this | study to evalua | ate the clinica |
| Denormance | | | |

| | Clinical Investigation Plan | | Page 9 of 2 |
|---|---|---|---|
| Cli | nical Investigation Plan: | Doc. No: | CIA No: 176 |
| | Hour Invocagation France | Revision: | В |
| . Lite | erature Review | | |
| structive | sleep apnea (OSA) is a prevalent health issue in western world | d effecting 24 | 1% of men ar |
| charact | en of the middle age population, and affecting around 2-4% of the crized by periodic collapse of the upper airway during sleep. CP. | AP is the pri | nary treatme |
| oatients | with OSA <sup>3,4</sup> . | ' | |
| Pre | olimical Tooting | | |
| Pre | clinical Testing | | |
| Pre | vious Clinical Experience | | |

| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inc | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIV | vestigation Fian. | Revision: | В |

| | Clinical Investigation Plan: | | |
|---|---|---|---|
| | Chinton in Conguine Film | Revision: | В |
| 7.5. | Justification for Administration | | |
| | | rial have be | en previously |
| testec | | | |
| 8. | Objectives of the Clinical Investigation | | |
| 8.1. | <u>Hyp</u> othesis | | J P . J. 990 |
| The | investigational device clinical performance will be acceptable in t | erms of pro | duct reliability, |
| шетар | by effectiveness and user feedback. | | |
| 8.2. | Objectives | | |
| 0.2. | Objectives | | |
| The p | rimary objective for this investigation is to evaluate whether the investig | ational dev | ice treats the |
| | ipant safely, effectively and reliably | , | |
| | econdary outcome of this investigation is the participant perception of the | he device th | rough the |
| partic | ipant perception questionnaire, | | |
| 0 2 | Population | | |
| 8.3. | Population | h a diagnaa | : |

This investigation will include a total of 150 adult participants (22 or older) with a diagnosis of OSA and a PAP (CPAP or AutoCPAP) prescription. They may be either experienced users of PAP or naïve to PAP therapy. Further details are included in Section 9.8 Inclusion/Exclusion Criteria.

### 8.4. Risks

Positive airway pressure therapy is considered to be the gold-standard therapy for individuals with OSA (Section 7.2). The treatment is considered to be extremely safe and any adverse effects are usually short term and easily resolvable. Adverse effects can be caused by an ill-fitting mask, too much or too little pressure being delivered to the participant, existing or developing nasal congestion during CPAP use. Individuals that are contraindicated for CPAP therapy will be excluded during screening. For more information on contraindications, warnings and precautions refer to the user manuals provided in CIA-176,

The primary risk within the scope of this study that the pressure may be slightly too high or slightly too low

| Fishe | &Paykel FHCARE Clinical Investigation Plan | | |
|---|---|---|---|
| | Clinical Investigation Plan: | Doc. No: | CIA No: 176 |
| | | Revision: | В |
| is too | In the case of the pressure being eutic), this may result in the participant having sleep disordered breathingh, then the participant may be uncomfortable during CPAP use. Eith articipant feeling more tired than usual the next day. Other risks side effects of CPAP related to nasal these risks are common to CPAP devices, and this study in the case of the pressure being eutic). | ng events.<br>her of these<br>dryness ar | If the pressure e may result in and congestion. |
| | sual therapy. | <b>Op. 300</b> | g. cattor |
| 8.5. | Essential Requirements of the Relevant Directive | | |
| | Clinical Investigation Design Type of Investigation an open-label (investigators and participants are un-blinded and informal) single arm study. The intended treatment will not | ned of inter<br>ot be rando | |
| 9.2. | Controls | | |
| | ntrol group will be used in this study | | |
| 9.3. | Bias | | |
| Partic | pants will not be blinded to any therapy settings for the duration of the | trial. | |
| | | | _ |
| 0.4 | End Points | | |
| 9.4. | | | |
| | <b>Primary Outcomes</b> rimary outcomes of effectiveness, safety and reliability will be measured | d by: | |
| 9.4.2. | Secondary Outcomes | | |
| The s | econdary outcome of this investigation is the participant perception of the | ne device | |
| _ | | | |
| 9.5.<br>The fo | Variables llowing variables will be recorded during the investigation: | | |

| Fisher & Paykel<br>HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inv | estigation Plan: | Doc. No: | CIA No: 176 |
| Cillical Iliv | estigation Fian. | Revision: | В |



### 9.6. Measurements

The following measurements will be performed during the study



# 9.7. Equipment

Each participant will be issued the following:



### 9.8. Inclusion / Exclusion criteria

The inclusion criteria for participants in this investigation will be:

- Aged 22 and over (FDA defined as adult).
- Diagnosed with OSA by a practicing physician and prescribed PAP (CPAP or AutoCPAP) therapy.

| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inv | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cililical IIIV | estigation Fian. | Revision: | В |

- For experienced users of PAP (CPAP or AutoCPAP):
  - Using the PAP of more than 4 hours/night for 70% during the last 30 days (justification allowed by the investigator of each site if the participant does not meet this compliance but is deemed suitable for this trial).

The exclusion criteria for participants in this investigation will be:

- Contraindicated for PAP (CPAP or AutoCPAP) therapy.
- Persons with other significant sleep disorder(s) (e.g. periodic leg movements, insomnia, central sleep apnea).
- Persons with obesity hypoventilation syndrome or congestive heart failure.
- Persons that require supplemental oxygen with their PAP (CPAP or AutoCPAP) device.
- Persons with implanted electronic medical devices (e.g. cardiac pacemakers).
- Persons who are pregnant or think they might be pregnant.
- Persons whose is not fluent in spoken and written English.

### 9.9. Point of Enrolment

A participant shall be considered enrolled into the investigation once they have been screened for the inclusion/exclusion criteria, signed the informed consent form and taken the device home to use for the first time.

# 9.10. Patient Procedure

| Fisher & Paykel<br>HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inv | estigation Plan: | Doc. No: | CIA No: 176 |
| Cillical Iliv | estigation Flan. | Revision: | В |



### 9.11. Withdrawal Criteria

Participants enrolled in this investigation will be notified that they have the right to withdraw from the investigation at any time, without prejudice to their medical care and are not obliged to state their reasons. The investigator will follow-up any withdrawals.

Additionally, the investigator may withdraw a participant at any time for the following reasons:

- 1. Inability to tolerate trial PAP device due to nasal obstruction or claustrophobia
- 2. Protocol violation
- 3. Serious illness
- 4. Adverse events

The reason for participant discontinuation in the investigation is to be recorded in the CRF and will be included in any clinical investigation report.

| Fisher&Paykel | Clinical Investigation Plan | | |
|---------------|-----------------------------|-----------|---------------|
| Clinical Inv | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIv | estigation Flan. | Revision: | В |

| 9.12. Number of Trial Subjects 150 trial participants will be included in this investigation, |
|---|
| 9.13. Follow up Plan |
| Participants remain under the medical care of their usual care provider during the trial, and after the trial has concluded. |
| 9.14. Foreseeable Complications PAP use may irritate certain conditions and may be temporarily contraindicated in participants who exhibit sinus infection, middle ear infection or a perforated ear drum. Participants that are contraindicated for PAP will be excluded from the investigation. |
| The participant will be instructed to cease using the device if they think the device is malfunctioning, not treating them or if they feel uncomfortable using the device; and that they should immediately swap to their usual PAP device (if available) for the rest of the night and contact a member of the research team as soon as possible. The research team will then assess with the participant if the problem can be resolved, or withdraw them from the trial. |
| <ul> <li>10. Clinical Trial Documentation</li> <li>10.1. Consent and Recruitment</li> <li>Informed consent will be taken for all participants enrolled in this investigation. A copy of the information sheet and consent form is included with the ethics application,</li> </ul> |
| 10.2. Case Report Form Investigation data will be recorded in source documents and attached to the Case Report Form (CRF) for both the administration of the investigation and collection of participant data. |
| 10.2.1. Case Report Form Signatories Case Report Form Signatories will be included on the Delegation of Authority in the site regulatory file. |
| 10.3. Insurance Statement A copy of the insurance statement will be included in the CIA folder |

| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inv | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIV | vestigation Fian. | Revision: | В |

### 10.4. Record of Deviations



| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inc | vestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIV | vestigation Fian. | Revision: | В |

### 10.8. Statistical Termination

There is no criteria for statistical termination for this investigation.

### 10.9. Statistical Procedure Deviations

There is no criteria for statistical procedure deviations for this investigation.



10.11. Statistical Data Management



### 11. Adverse Events and Termination

# 11.1. Emergency Contact Details

The participant will contact their following investigator if there are any adverse events:

Name: Matt Uhles

Address: Clayton Sleep Institute, Email: uhlesm@claytonsleep.com

Phone: 314-645-6005



| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical In | evestigation Plan: | Doc. No: | CIA No: 176 |
| Cillical III | vestigation Fian. | Revision: | В |

### 11.2. Foreseeable Adverse Events

Foreseeable adverse events for this investigation include the following:

These foreseeable adverse events are the same as those for a PAP patient on their usual therapy.

11.3. Reporting Adverse Events

### 11.4. Early Termination

If a participant is struggling with therapy during the investigation and we are unable to resolve the issue causing the problem, the participant may be terminated early from the investigation. The participant also has the right to withdraw from the investigation at any point without a need for a reason.

If \_\_\_\_\_\_ it becomes clear that the \_\_\_\_\_ device is not treating participants effectively, the investigator may terminate the trial in its entirety.

The following documentation is required if the appropriate party terminates a clinical trial.

### 11.4.1. Investigator

If the investigator terminates or suspends a trial without prior agreement of the sponsor, the investigator should inform the institution, where required by the applicable regulatory requirements and the

| Fisher & Paykel HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Investigation Plan: | | Doc. No: | CIA No: 176 |
| | | Revision: | В |

investigator/institution should promptly inform the sponsor and the IRB, and should provide the sponsor and the IRB a detailed written explanation of the termination or suspension.

### 11.4.2. **Sponsor**

If the sponsor terminates or suspends a trial, the investigator should promptly inform the institution, where required by the applicable regulatory requirements, and the investigator/institution should promptly inform the IRB and provide the IRB a detailed written explanation of the termination or suspension.

### 11.4.3. Institutional Review Board (IRB)

If the IRB terminates or suspends its approval/favorable opinion of a trial the investigator should inform the institution, where required by the applicable regulatory requirements, and the investigator/institution should promptly notify the sponsor and provide the sponsor with a detailed written explanation of the termination or suspension.

| 12. | Publication Policy |
|-----|--------------------|

## 13. Approval

Signing the below approval indicates that the principal investigator(s) (PI) in each trial center and the sponsor agree to this version of Clinical Investigator Plan.

| Principal Investigator Approval: PI Name: |
|-------------------------------------------|
| PI Signature: |
| Date (dd/mmm/yyy): |
| Sponsor Approval Sponsor Name: |
| Sponsor Signature: |
| Date (dd/mmm/yyy): |

### 14. References

| Fisher & Paykel<br>HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Investigation Plan: | | Doc. No: | CIA No: 176 |
| | | Revision: | В |



| Fisher & Paykel<br>HEALTHCARE | Clinical Investigation Plan | | |
|---|---|---|---|
| Clinical Inv | restigation Plan: | Doc. No: | CIA No: 176 |
| Cillical IIIV | estigation Fian. | Revision: | В |

| Fisher & Paykel | Clinical Investigation Plan | | | |
|---|---|---|---|---|
| Clinical Inv | restigation Plan: | Doc. | No: | CIA No: 176 |
| Cimical inv | estigation Fian. | Revis | sion: | В |